CLINICAL TRIAL: NCT02600286
Title: LONG-TERM EFFECTS TOLERANCE AND THE Ulipristal Acetate IN DISEASE Charcot-MARIE-TOOTH TYPE OF 1A
Brief Title: Ulipristal Acetate In Disease Charcot-Marie-Tooth Type of 1A
Acronym: UPACOMT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6100
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: CMT1A
Keywords: Physical medicine and rehabilitation; Neurology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Arm (1) will be randomised to receive either :
  * 5 mg/per os of EllaOne every day through 12 months.
  * 10 mg/per os of EllaOne every day through 12 months.
  * EllaOne placebo/per os every day through 12 months.
  Interventions: Drug: EllaOne; Drug: EllaOne placebo
- 2 (Experimental): Arm (2) will be randomised to receive either :
  * 5 mg/per os of EllaOne every day through 12 months.
  * 10 mg/per os of EllaOne every day through 12 months.
  * EllaOne placebo/per os every day through 12 months.
  Interventions: Drug: EllaOne; Drug: EllaOne placebo
- 3 (Experimental): Arm (3) will be randomised to receive either :
  * 5 mg/per os of EllaOne every day through 12 months.
  * 10 mg/per os of EllaOne every day through 12 months.
  * EllaOne placebo/per os every day through 12 months.
  Interventions: Drug: EllaOne; Drug: EllaOne placebo

INTERVENTIONS:
Drug: EllaOne — * 5 mg/per os of EllaOne every day through 12 months.
  * 10 mg/per os of EllaOne every day through 12 months.
  * EllaOne placebo/per os every day through 12 months.
  Other Names: 1: Experimental; 2: Experimental; 3: Experimental
Drug: EllaOne placebo — * 5 mg/per os of EllaOne every day through 12 months.
  * 10 mg/per os of EllaOne every day through 12 months.
  * EllaOne placebo/per os every day through 12 months.
  Other Names: 1: Experimental; 2: Experimental; 3: Experimental

SUMMARY:
The disease Charcot-Marie-Tooth disease type 1A (CMT1A) is the most common inherited peripheral neuropathy, for which no treatment has proved its effectiveness. It is autosomal dominant, associated with a duplication of the chromosome 17p11.2 region which leads to overexpression of the gene and the protein-peripheral myelin protein-22 (PMP22), a major component of peripheral myelin.

In animals and humans, PMP22 mRNA level of glutathione S-transferase theta 2 and Cathepsin A (markers of oxidative stress), detected in a skin biopsy are markers that may play a role in the prognosis evolution of the disease. Furthermore, several studies have shown that the administration of progesterone increased the expression of PMP22 gene (measured in a skin biopsy) and worsening symptoms. In contrast, anti-progestins reduce the synthesis of PMP22 and improve symptoms in rat CMT1A.

The long-term safety of anti-progesterone was evaluated for mifepristone (RU486) ulipristal acetate and (EllaOne®). Few side effects have been reported including a few cases of endometrial hyperplasia reversible upon discontinuation of treatment. With the RU486, rare cases of adrenal androgen and failure have been observed. However, EllaOne® has low antagonistic action on the glucocorticoid receptor and no action on androgen receptors. The investigators therefore believe that it will be well tolerated in humans and will reduce the synthesis of PMP22 and the action of oxidative stress by improving disability of patients.

ELIGIBILITY:
Inclusion Criteria:

* Male 18-70 years
* CMT1A proven genetically (17p11.2 duplication)
* symptomatic CMT1A (MRC score <5 in at least one muscle group)
* Non severe axonal impairment (amplitude of the motor evoked potential on the median nerve and / or ulnar than 50% of normal)
* Subject contacted with a valid phone number
* Subject affiliated to a social security scheme
* Subject has been informed of the results of the medical examination prior

Exclusion Criteria:

* Another cause of neuropathy: Chronic alcohol intoxication, chemotherapy, diabetes, kidney failure, monoclonal gammopathy, cryoglobulin, B12 deficiency, hepatitis B / C, HIV, Lyme or poliomyelitis
* Liver failure
* Lapp lactase deficiency, malabsoprtion syndrome glucose / galactose
* Support long-term drug interacting with the CYP3A4
* Patients with indication against xylocaine adrenaline
* In the biopsy site: surgery, skin disease or local infection
* Immunosuppression innate or acquired
* Hypersensitivity to the active substance / excipient
* uncontrolled severe asthma
* Treatment with vitamin C or vitamin B3 in the four weeks preceding randomization
* Orthopaedic surgery of the lower limbs in the 6 months prior to randomization or planned
* Against indication xylocaine adrenaline
* Malfunction of the innate or acquired coagulation

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Analysis of the effectiveness of Ellaone. This will be assessed by the production of RNA PMP22 using skin biopsy. | 12 months after treatment with EllaOne

CONTACTS AND LOCATIONS:
Overall Officials: Andoni Echaniz-Laguna, MD, Study Director — University Hospital, Strasbourg, France; Nicolas Collongues, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (5):
- France (5):
  - Service d'Explorations et pathologies neuro- musculaires, Besançon
  - Département de Neurologie, Dijon
  - Département de Neurologie, Nancy
  - Unité de pathologie neuro-musculaire, Paris
  - Département de Neurologie Centre de Référence des Maladies Neuromusculaires Grand Est (CERNEST) Hôpital de Hautepierre, Strasbourg